CLINICAL TRIAL: NCT01004042
Title: Evaluation of Quality of Life and Self-esteem After Botulinum Toxin type-a (Botox®) Injections in Depressed and Non-depressed Patients
Brief Title: Quality of Life and Self-esteem After Botox® Injections in Depressed and Non-depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-CBED09-02
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Depression; Quality of Life
Keywords: Depression; Botulinum toxin; Glabella; Quality of life; Self-steem
MeSH Terms: conditions — Depression | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed subjects (Active Comparator): Diagnosis of depression (diagnostic criteria from DSM-IV-TR and MINI International Neuropsychiatric Interview - Brazilian version 5.0.)They must be using a therapeutic dose of antidepressant for at least 2 months before the intervention prescribed by a psychiatrist.
  Interventions: Drug: Botulinum Toxin Type A
- Non Depressed subjects (Active Comparator): Subjects with no diagnosis of depression
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Subjects included in the study will receive injections of 20 U (as minimal dose) to 40 U (as maximum dose) of BTX-A (BOTOX®/Allergan, USA) diluted in 0.9% saline, according to standard injections of 4U in 5 points of glabellar area as the treatment.
  Other Names: Botox®

SUMMARY:
The primary objective of this study is to determine the alterations in quality of life and self-esteem after BOTOX® injections in the glabella in depressed and non-depressed patients.

The secondary objective of this study are:

* to assess wrinkles improvement
* to evaluate depressive symptoms using Beck Depression Inventory before and after Botox® injections.
* to elucidate that depression is not a contraindication for botulinum toxin injections.

DETAILED DESCRIPTION:
The study consists of two groups: one with diagnosis of depression (diagnostic criteria from DSM-IV-TR and MINI International Neuropsychiatric Interview - Brazilian version 5.0) and other without diagnosis of depression.

Subjects with depression will be part of group 1. They must be using a therapeutic dose of antidepressant for at least 2 months before the intervention prescribed by a psychiatrist.

Subjects with no diagnosis of depression will be part of group 2. Subjects included in the study will receive injections of 20 U (as minimal dose) to 40 U (as maximum dose) of BTX-A (BOTOX®, Allergan, USA) diluted in 0.9% saline, according to standard injections of 4U in 5 points of glabellar area as the treatment.

Four visits will be scheduled. Visit 0 (baseline), Visit 1 (intervention), visit 2 (4 weeks), visit 3 (8 weeks) visit 4 (12 weeks).

The scales for the assessment of depressive symptoms, Beck Depression Inventory (BDI), will be applied at visits 1,2,3,4; WHOQOL BREF will be applied at baseline visit and 4.

Rosenberg Self-Esteem Scale will be applied in all visits. Photographs will be taken as well as the dermatological evaluation of the wrinkles and folds will be assessed using a 4-points validated Severity Wrinkles Scale, and psychiatric evaluation as well, in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects,aged between 25 to 60 years;
2. Subjects diagnosed as having major depression according to the criteria of DSM-IV, MINI International Neuropsychiatric Interview (MINI Brazilian version 5.0.0);
3. Subjects who are being administered a therapeutic dose of an approved, prescribed antidepressant medication (pattern doses of the literature), and have been using mentioned medication at a stable therapeutic dose for at least three months prior to the randomization visit;
4. Subjects with mild (1), moderate (2) or severe (3) glabellar frown lines while at rest according the Severity Wrinkles Scales;
5. Female subjects of childbearing age that present a negative urine pregnancy test and are using an effective contraceptive method;
6. Subjects who had never received botulinum toxin A previously;
7. Subjects agreeing to take part of the study, after being fully informed of the purpose and the nature of the investigation and after having signed the informed consent form;
8. Subjects who will be available throughout the duration of the study;
9. Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol;
10. Subjects with Critical appreciation preserved, attested by their assistant psychiatrist (for group1);
11. Subjects who reside with other family members who assume co-responsibility in the study.

Exclusion Criteria:

1. Subjects whose medical history and physical examination present clinical pathology, as myasthenia gravis, Eaton-Lambert Syndrome, neoplasm, muscular diseases, motor neuron diseases, systemic autoimmune or neurological diseases;
2. Pregnant or women in breastfeeding, or women planning to become pregnant
3. Subjects with suicide risk;
4. Subjects addicted to alcohol or illegal drugs within the last 6 months;
5. Subjects using amino glycoside and penicillamine antibiotics, quinine and Ca2+ channel blockers;
6. Subjects using medications that, in the opinion of the investigator may cause depression, such as beta-blockers, oral corticosteroids and interferon;
7. Subjects who, in the opinion of the investigator, may potentially require psychiatric hospitalization during the course of the study;
8. Subjects with inflammation or active infection in the area to be injected;
9. Subjects with a history of non-adherence to medical treatment, or who demonstrate unwillingness to adhere to the study protocol;
10. The presence of any additional active DSM-IV Axis I diagnosis, or mental retardation;
11. History of psychiatric hospitalization within the past three years.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator — Brazilian Center For Studies in Dermatology
Locations (1):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depressed Subjects | Non Depressed Subjects
Started | 25 | 25
Completed | 21 | 25
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depressed Subjects | Non Depressed Subjects | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7) | 48 (7) | 49 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Measure Description: Phototype I - Pale white skin, blue/green eyes, blond/red hair; Always burns, does not tan Phototype II - Fair skin, blue eyes; Burns easily, tans poorly Phototype III - Darker white skin; Tans after initial burn Phototype IV - Light brown skin; Burns minimally, tans easily Phototype V - Brown skin; Rarely burns, tans darkly easily Phototype VI - Dark brown or black skin; Never burns, always tans darkly
  Participants
    Fitzpatrick Skin Phototype I: Phototype I | 0 | 0 | 0
    Fitzpatrick Skin Phototype I: Phototype II | 7 | 3 | 10
    Fitzpatrick Skin Phototype I: Phototype III | 15 | 21 | 36
    Fitzpatrick Skin Phototype I: Phototype IV | 2 | 1 | 3
    Fitzpatrick Skin Phototype I: Phototype V | 1 | 0 | 1
    Fitzpatrick Skin Phototype I: Phototype VI | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 25 | 25 | 50
Marital status [Count of Participants; unit: Participants]
  Married or steady relationship | 14 | 13 | 27
  Single | 3 | 4 | 7
  Divorced | 8 | 8 | 16
Education [Count of Participants; unit: Participants]
  College | 11 | 9 | 20
  College (not completed) | 2 | 4 | 6
  High School | 12 | 10 | 22
  Middle School | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rosenberg Self-Esteem Scale
Description: Measure of self esteem for research purposes.
  Ten questions graded from 0 to 3 as described below:
  Questions 1, 3, 4, 7, 10
  0 - Totally agree
  1. - Agree
  2. - Disagree
  3. - Totally disagree
  Questions 2, 5, 6, 8, 9
  3 - Totally agree 2 - Agree
  1 - Disagree 0 - Totally disagree
  The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
Time Frame: Baseline, Day 1 (intervention), Week 4, Week 8, Week 12
Population: per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects | Non Depressed Subjects
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 13.9 (5.3) | 24.6 (4.3)
  Day 1 (intervention) | 13.5 (5.0) | 23.3 (5.3)
  Week 4 | 15.2 (5.8) | 23.5 (4.9)
  Week 8 | 17.1 (5.9) | 24.4 (4.6)
  Week 12 | 16.9 (6.5) | 24.2 (4.9)

2. Primary Outcome: Beck Depression Inventory (BDI)
Description: BDI is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Each question is graded from 0 to 3.
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Time Frame: Baseline, Day 1 (intervention), Week 4, Week 8, Week 12
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects | Non Depressed Subjects
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 27.4 (5.2) | 6.7 (5.5)
  Day 1 (intervention) | 24.3 (8.8) | 5.8 (4.5)
  Week 4 | 17.0 (7.9) | 5.3 (4.1)
  Week 8 | 14.9 (9.9) | 4.5 (4.4)
  Week 12 | 12.5 (7.9) | 4.0 (3.4)

3. Secondary Outcome: WHOQOL-BREF
Description: The WHOQOL-BREF is a scale for the quality of life assessment developed by the World Health Organization. It is composed by 26 questions graded from 1 to 5.
  Scoring:
  1 to 2.9 - needs improvement 3 to 3.9 - regular 4 to 4.9 - good 5 - very good
  Question 1 asks about the individual's overall perception of quality of life. Results refer to question 1.
Time Frame: Baseline, Day 1 (intervention), Week 4, Week 8, Week 12
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects | Non Depressed Subjects
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 2.9 (0.77) | 3.9 (0.49)
  Day 1 (intervention) | 2.9 (0.85) | 4.0 (0.81)
  Week 4 | 3.6 (0.60) | 4.1 (0.53)
  Week 8 | 3.5 (0.89) | 4.1 (0.57)
  Week 12 | 3.4 (0.81) | 4.1 (0.57)

4. Secondary Outcome: Wrinkle Severity Scale (WSS) at Rest
Description: The injection of botulinum toxin type A causes muscle paralysis, reducing facial lines. Wrinkle scales are used to grade the muscular effects of botulinum toxin.
  The WSS is a 4-point validated scale for forehead lines:
  0 - None
  1. - Mild
  2. - Moderate
  3. - Severe
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects | Non Depressed Subjects
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 1.6 (0.76) | 1.5 (0.51)
  Week 4 | 0.4 (0.61) | 0.5 (0.59)
  Week 8 | 0.4 (0.62) | 0.4 (0.58)
  Week 12 | 0.4 (0.62) | 0.7 (0.58)

5. Secondary Outcome: Wrinkle Severity Scale (WSS) at Maximum Contraction
Description: as for outcome 4
Time Frame: Baseline, Day 1 (intervention), Week 4, Week 8, Week 12
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects | Non Depressed Subjects
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 2.6 (0.69) | 2.7 (0.48)
  Week 4 | 1.1 (0.64) | 1.2 (0.65)
  Week 8 | 0.9 (0.80) | 1.2 (0.80)
  Week 12 | 1.4 (0.70) | 1.7 (0.56)

ADVERSE EVENTS:
Arm/Group | Depressed Subjects | Non Depressed Subjects
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depressed Subjects (N=25) | Non Depressed Subjects (N=25)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Edema on the nose and infraorbital region. Patient with past history of latex allergy.
Mild eyebrow ptosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild ptosis in medial third of the right eyebrow

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes